CLINICAL TRIAL: NCT06784908
Title: Stress-immune Mechanisms for People Living With HIV, CUD and Depression
Brief Title: Stress and Pain in People Living With HIV
Acronym: HIV Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000038503; 1R01DA061995-01 (NIH)
Record Dates: First submitted 2025-01-16; First posted 2025-01-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: HIV; Depression; Cannabis Use Disorder; Stress; Pain
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIV-positive (PLWH+) (Experimental): Participants that are HIV-positive only will undergo 2 Within Subjects factors of Condition, Stress and No Stress (order of condition randomly assigned and counterbalanced)
  Interventions: Other: Yale Pain Stress Task (YPST)
- HIV-positive and complex morbidity (PLWH/CM+) (Experimental): Participants that are HIV-positive with complex morbidities will undergo 2 Within Subjects factors of Condition, Stress and No Stress (order of condition randomly assigned and counterbalanced)
  Interventions: Other: Yale Pain Stress Task (YPST)
- Healthy control (HC) (Experimental): Participants that are not HIV-positive and no complex morbidities will undergo 2 Within Subjects factors of Condition, Stress and No Stress (order of condition randomly assigned and counterbalanced)
  Interventions: Other: Yale Pain Stress Task (YPST)
- Control and complex morbidity (HC+CM) (Experimental): Participants that are not HIV-positive and have complex morbidities will undergo 2 Within Subjects factors of Condition, Stress and No Stress (order of condition randomly assigned and counterbalanced)
  Interventions: Other: Yale Pain Stress Task (YPST)

INTERVENTIONS:
Other: Yale Pain Stress Task (YPST) — Individuals in the experimental cohort will be scheduled for 2 experimental sessions 1-3 days apart. The YPST stress experiment includes a stress and no-stress session (order randomly assigned, counter-balanced across subjects), and involves multiple (up to 3) unpredictable number of consecutive 3-minute trials of ice-bath (stress) or warm-bath (no stress) forearm immersion (stress) with subjective, physiologic endocrine and immune assessments repeated at specified time points.

SUMMARY:
This is a basic human experimental study utilizing 4 groups of individuals with and without HIV and complex morbidities of cannabis use disorder and major depression who will participate in 2 sessions of the Yale Pain Stress Task (YPST) and follow-up phase to assess drug use and mood symptoms.

DETAILED DESCRIPTION:
This study aims to address research gaps using a powerful and novel cross-diagnostic approach with multiple complementary approaches to examine the overarching hypothesis that PLWH+CM exhibit impaired stress-related HPA and HPA-immune function due to alterations in epigenetic mechanisms, and these stress-related HPA-immune and related epigenetic aberrations predict distress, craving and substance use symptoms underlying PLWH complex morbidities. This hypothesis will be tested using a combined human experimental stress challenge approach with prospective longitudinal assessment of daily distress, and substance use symptoms as well as assessment of chronic stress (C-stress), social determinants of health (SDoH), and resilience in experimental cohorts of PLWH with and without CM and those without HIV with and without CM.

ELIGIBILITY:
Inclusion Criteria:

* good health as verified by screening examination
* Able to read English and complete study evaluations and provide informed written and verbal consent. Additional criteria PLWH
* HIV-1 lab test positive
* undetectable viral load
* good ART adherence

Additional criteria by group:

PLWH +CM:

* CB positive urine toxicology
* meet DSM-5 criteria for CUD and MDD as assessed using SCID-I. HC
* HIV-1 test negative
* urine toxicology negative
* no major medical and psychiatric diagnoses based on DSM-V.

PLWH Only:

* HIV-1 test positive
* urine toxicology negative
* no major medical and psychiatric diagnoses based on DSM-V.

CM Only:

* HIV-1 test negative
* urine toxicology positive
* meet DSM-5 criteria for CUD and MDD as assessed using SCID-I

Exclusion Criteria:

* meet primary, current moderate and severe criteria for other SUD including cocaine, alcohol, opiates, sedatives, nicotine
* current use or past history of cocaine or opioid use disorder
* history of any psychotic disorder
* current diagnoses of bipolar disorder and PTSD
* psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania)
* significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology that would interfere with study participation
* medications with known central effects on HPA axis and cytokines/immune function
* women who are pregnant, nursing or those using hormonal birth control that affect HPA axis cortisol responses.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in cortisol levels | day 1 and day 3
  Mean change in cortisol levels (pg/ml) assessed using repeated blood sampling over 2 hour period on 2 separate days to extract plasma for cortisol measurement using standard RIA assay procedures.
Change in adrenocorticotropic hormone (ACTH) levels | day 1 and day 3
  Mean change in pain stress assessed using repeated blood sampling over 2 hour period on 2 separate days to extract plasma for ACTH measurement using standard RIA assay procedures.
Change in pain stress | day 1 and day 3
  Mean change in pain stress assessed using repeated sampling over 2 hour period on 2 separate days using 10-point visual analog scales (VAS) where 0 is not at all and 10 is the most pain being experienced.

SECONDARY OUTCOMES:
Mean behavioral pain tolerance | day 1 or day 3
  Time in seconds that hand remains immersed in ice cold and warm water over 3 trials of 3 minutes each as a measure of behavioral pain tolerance
Mean Heart Rate | day 1 and day 3
  Heart rate (bpm) assessed using repeated sampling over 2 hour period on 2 separate days using standard heart rate monitor.
Mean Blood pressure (systolic and diastolic) | day 1 and day 3
  Blood pressure (mmHg), systolic and diastolic,assessed using repeated sampling over 2 hour period on 2 separate days using standard blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, Ph.D., Principal Investigator — Yale University
Locations (1):
- The Yale Stress Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified data will be uploaded into National Institute of Mental Health Data Archive (NDA) data repository.